CLINICAL TRIAL: NCT01979991
Title: Model-Based Image Reconstruction for X-Ray CT in Lung Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); General Electric (Industry)
Responsible Party: Principal Investigator, Jeffrey Fessler PhD., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00038447
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT Imaging and Reconstruction (Experimental): To develop a MBIR (model-based image reconstruction) method that will improve X-ray CT lung imaging by improving image quality and reducing dose.
  Interventions: Procedure: CT Imaging and Reconstruction

INTERVENTIONS:
Procedure: CT Imaging and Reconstruction — Patients will be consented for their permission to save and use the sinogram from their CT chest/lung scan. The sinogram will be de-identified and sent to an archive system for storage.
  Later it will be exported to a computer for processing using MBIR (model based image reconstruction). The newly processed images will then be read by blinded readers. The quality of the images will be reviewed to determine if they are as readable and accurate as CT images created with the software that is currently being used.

SUMMARY:
To develop a computer program that will improve CT image quality and decrease the amount of x-ray radiation that future patients may be exposed to when they have a CT examination.

DETAILED DESCRIPTION:
We will be asking patients for their permission to save and use the sinogram from their CT scan. The sinogram will be de-identified and sent to an archive system for storage. It will be exported to a computer for processing using MBIR (model based iterative reconstruction). MBIR (model based iterative reconstruction) is a new method being developed to process CT sinograms. The newly reconstructed images will be reviewed by experts to determine if they are as readable and accurate as CT images created with the software that is currently being used. Sinogram data and the reconstructed images will be shared with collaborating researchers at General Electric Global Research.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older 2. No medical or psychiatric condition precluding informed consent

-

Exclusion Criteria:

1. Inability to lie flat on the back with arms raised over the head for 30min.
2. Metallic implants or metallic devices in the chest or back.
3. Participation in other research trials involving ionizing radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2010-08; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Developement of a computer program to improve CT image quality | 6 years
  Sinograms will be retrieved by an archive system and processed by MBIR (model-based image reconstruction) methods that we are developing that improve image quality (reduce noise, improve spatial resolution, reduce artifacts). We will evaluate the image quality both quantitatively and qualitatively.
  We hope to develop and benchmark methods for algorithm acceleration to enable routine clinical use of MBIR (model-based image reconstruction) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fessler, PhD, Principal Investigator — University of Michigan Hospital; Jeffrey Fessler, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States